CLINICAL TRIAL: NCT04125303
Title: The Effectiveness of a Brief Motivational Nursing Intervention to Reduce Psychoactive Substance Consumption in Entertainment-sector Workers: A Transversal, Observation, and Semi-experimental Study
Brief Title: The Effectiveness of a Brief Motivational Nursing Intervention
Acronym: BMNI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Isabel Almodóvar Fernández, Nursing Coordinator, Cardenal Herrera University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DGNRI316-06-23
Record Dates: First submitted 2019-09-30; First posted 2019-10-14 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Behavior, Addictive
Keywords: cannabis; cocaine; alcohol; entertainment workers; nursing interventions
MeSH Terms: conditions — Behavior, Addictive; Marijuana Abuse

STUDY DESIGN:
Masking Description: Outcomes assesor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Based on NANDA diagnosis recommendations, entertainment-sector workers were asked to record their perceptions and the meaning of their substance-use problem in a diary. The intervention was subsequently designed based on brief motivational psychoeducational therapy (BMPT).
  Interventions: Behavioral: brief motivational psychoeducational therapy

INTERVENTIONS:
Behavioral: brief motivational psychoeducational therapy — The brief motivational psychoeducational therapy (BMPT) it lasted an average of 90 min and followed the following structure: (i) brainstorming the concepts of health, lifestyle, and substance-use prevention; (ii) analysis of a work accident at an international rock group concert, which was used to generate (iii), a debate on consumer habits (30 min); (iv) discussion of the substance types and classifications known by the participants; (v) Prochaska and DiClemente's stages of change and (vi), the consequences of drug use (50 min); and finally, (vii) a true/false quiz used to discuss myths and beliefs about drugs (10 min).

SUMMARY:
This was a two-staged study undertaken in entertainment-sector workers in Spain: the first part was transversal and observational, and the second was semi-experimental. A short group-based motivational intervention session was implemented by nursing staff, and a before and after evaluation was completed. By reducing the patients' perception of their quality of life, this brief nursing intervention facilitated a favourable increase in the motivation for change among these workers and was effective in 12% of cases.

DETAILED DESCRIPTION:
Checking whether changes in the perception of the quality of life related to health, after the nursing intervention, influence these patients' motivation to change. This was a two-staged study undertaken in entertainment-sector workers in Spain: the first part was transversal and observational, and the second was semi-experimental. First part undertook in 284 entertainmentsector workers, selected by non-probabilistic sampling, while second part undertook in 50 entertainment-business workers, selected by consecutive sampling from those who consumed substances. A short group-based motivational intervention session was implemented by nursing staff, and a before and after evaluation was completed. The EuroQol-5D and Test for the Evaluation of the Quality of Life in Addicts to Psychoactive Substances (TECVASP) were used. The patients' motivation to change was evaluated through the Stages of Change Readiness and Treatment Eagerness Scale.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years
* working conditions that fulfilled the Health and Safety requirements
* acceptance of the informed consent to participation.
* Drugs and alcohol users

Exclusion Criteria:

* younger than 18 or older than 65
* Non drugs and alcohol users

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
General perception of health related quality of life EQ-5D-3L | At 1 month
  Health related quality of life (HRQL) meassured by EQ-5D (EuroQuol) The EQ-5D-3L descriptive system comprises the following 5 dimensions, each describing a different aspect of health: mobility, self-care, usual activities, pain/disconfort and anxiety/depression. Each dimension has 3 respnse levels of severity: no problems, some problems, extreme problems. The respondent is asked to indicate his/her health state by checking the box next to the most appropiate response level of each five dimensions.
Health related quality of life TECVASP | At 1 month
  Assessment of the Quality of Life in Psychoactive Substance Addicts Test TECVAS
  It consists of 22 items (18 positive and 4 negative [items 15, 19, 20 and 21]) with a graded response format of five alternatives. The response alternatives are coded with the following alternatives: a) in the positive items: nothing (5 points), little (4 points), sometimes (3 points), enough (2 points) and much (1 point); b) in the negative items: nothing (1 point), little (2 points), sometimes (3 points), enough (4 points) and much (5 points). Therefore, in each element, a higher score represents a more positive evaluation of the content, and in the test, a higher score represents a better HRQL.
Motivation to change | At 1 month
  Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES Scale) SOCRATES is an experimental instrument designed to assess readiness for change in alcohol and drugs abusers. The instrument yields three factorially-derived scale scores: Recognition (Re), Ambivalence (Am), and Taking Steps (Ts). It is a public domain instrument and may be used without special permission. The statements describes a way that the user might (or might not) feel about his/her drug use. For each statement, he/she has to circle one number from 1 to 5, to indicate how much they agree or disagree with it right now.

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Haro Cortés, Dr, Study Director — Universidad CEU cardenal Herrera-Consorcio Hospitalario Provincial de Castellón
Locations (1):
- University CEU Cardenal Herrera, Castellon, Castellón, Spain

REFERENCES:
- [Background] Almodovar-Fernandez I, Sanchez-Thevenet P, Benito A, Baquero A, Mari-Sanmillan MI, Haro G. The effectiveness of a brief motivational nursing intervention to reduce psychoactive substance consumption in entertainment-sector workers: A transversal, observation, and semi-experimental study. Int J Ment Health Nurs. 2019 Oct;28(5):1090-1098. doi: 10.1111/inm.12620. Epub 2019 Jun 11. PMID 31184429